CLINICAL TRIAL: NCT03164239
Title: The Effect of a Tailored Telephone and Email Based Physical Activity Intervention on Physical Fitness and Body Composition: a Randomized Controlled Trial
Brief Title: Aktiv i Sør: a Randomized Controlled Trial
Acronym: AiS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Agder (Other)
Collaborators: Norwegian School of Sport Sciences (Other)
Responsible Party: Principal Investigator, Monica Klungland Torstveit, Principal Investigator, University of Agder
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Aktiv i Sør
Record Dates: First submitted 2017-03-09; First posted 2017-05-23 (Actual); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group - telephone and print exercise intervention (Experimental): The intervention group (IG) received a total of three intervention packages, one every second month, during the intervention period. The first intervention package was distributed at intervention start. The intervention package consisted of a tailored exercise program, national recommendations for physical activity, prompts and reminders. Additionally the IG received fortnightly supportive motivational contact every two weeks, alternately by telephone og email
  Interventions: Behavioral: Intervention group - telephone and print exercise intervention
- Control group (No Intervention): The control group (CG) were encouraged to continue previous lifestyle.

INTERVENTIONS:
Behavioral: Intervention group - telephone and print exercise intervention — Intervention has previously been described.
  Arms: Intervention group - telephone and print exercise intervention

SUMMARY:
The purpose of this regional parallel-group RCT was to assess the effect of a six-month tailored telephone and email based physical activity intervention on various measures of physical fitness and body composition in a sample of physically inactive adults. A total of 111 physically inactive adults (40-55yr) from Agder, Norway were randomly allocated to either an intervention group (IG;n=56) or a no-intervention control group (CG;n=55). The IG received tailored exercise recommendations, every two months by email or mail (print) in addition to motivational follow-ups every second week, alternatively by email and telephone. Primary outcome measures were various objective measures of musculoskeletal and cardiorespiratory fitness in addition to various measures of body composition, including waist circumference, body mass index and fat percentage, which were assessed pre- and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

Participants were included in the study if they were

* healthy
* between the ages of 40-55
* residents of the Agder counties in Norway
* classified as physically inactive (not fulfill the recommendations for physical activity given by the Norwegian Directorate of Health
* within stage one to three of the five stages of change in the transtheoretical model stages of change

Exclusion Criteria:

Participants were excluded if they were

* Unhealthy/ill
* younger than 40 years or older than 55 years
* living outside the Agder counties in Norway
* allready fulfilling the national recommendations given by the Norwegian Directorate of Health
* within stage four or five of the five stages of change in the transtheoretical model stages of change

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 111 (Actual)
Dates: Start 2011-04-01 (Actual); Primary Completion 2011-10-01 (Actual); Study Completion 2012-02-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Cardiorespiratory fitness at 6 months | Data collected prior to (pre) and after (post) a 6 month intervention period. Pretest was conducted in March-April, 2011 and post test was conducted in October-November, 2011.
  Cardiorespiratory fitness was measured by a modified Balke protocol on a treadmill and registered in ml/kg/min
Change from Baseline Muscular endurance of the back extensors at 6 months | Data collected prior to (pre) and after (post) a 6 month intervention period. Pretest was conducted in March-April, 2011 and post test was conducted in October-November, 2011.
  The static back extension test recorded muscular endurance of the back extensors as number of seconds the subject managed to endure a static horizontal position, with their lower body supported by a bench (max 240 sec).
Change from Baseline Hand grip strength at 6 months | Data collected prior to (pre) and after (post) a 6 month intervention period. Pretest was conducted in March-April, 2011 and post test was conducted in October-November, 2011.
  Hand grip strength was registered to the nearest 1 kilogram (kg) using a hydraulic dynamometer
Change from Baseline Neuromotor fitness at 6 months | Data collected prior to (pre) and after (post) a 6 month intervention period. Pretest was conducted in March-April, 2011 and post test was conducted in October-November, 2011.
  Neuromotor fitness was registered using the one leg standing test where the duration each subject managed to hold a balancing position was recorded in seconds (max 60 seconds).
Change from Baseline Muscular dynamic endurance of and the ability to stabilize the upper body at 6 months | Data collected prior to (pre) and after (post) a 6 month intervention period. Pretest was conducted in March-April, 2011 and post test was conducted in October-November, 2011.
  Muscular dynamic endurance of and the ability to stabilize the upper body was registered using a modified push-ups test. The amount of correctly performed repetitions completed in 40 seconds, was recorded in number.
Change from Baseline Flexibility of the hamstring musculature at 6 months | Data collected prior to (pre) and after (post) a 6 month intervention period. Pretest was conducted in March-April, 2011 and post test was conducted in October-November, 2011.
  Flexibility of the hamstring musculature was recorded using the sit-and-reach test to the nearest half centimeter, using a specially designed box.
Change from Baseline Flexibility in the shoulder joint at 6 months | Data collected prior to (pre) and after (post) a 6 month intervention period. Pretest was conducted in March-April, 2011 and post test was conducted in October-November, 2011.
  Flexibility of the shoulder joint was registered to the nearest centimeter, using the back-scratch test. The mean registered flexibility score of both shoulders was recorded.
Change from Baseline Explosive power in the lower extremities at 6 months | Data collected prior to (pre) and after (post) a 6 month intervention period. Pretest was conducted in March-April, 2011 and post test was conducted in October-November, 2011.
  Explosive power in the lower extremities was recorded to the nearest centimeter, using the vertical jump test.
Change from Baseline Body mass index at 6 months | Data collected prior to (pre) and after (post) a 6 month intervention period. Pretest was conducted in March-April, 2011 and post test was conducted in October-November, 2011.
  Body mass index was calculated using the formula weight/height^2. Height and weight were measured using a measuring band (meters) and a weight scale (kilograms) respectively.
Change from Baseline Waist circumference at 6 months | Data collected prior to (pre) and after (post) a 6 month intervention period. Pretest was conducted in March-April, 2011 and post test was conducted in October-November, 2011.
  Waist circumference was registered using a measuring band and the mean of two measures was recorded to the nearest half-centimeter.
Change from Baseline Fat percentage at 6 months | Data collected prior to (pre) and after (post) a 6 month intervention period. Pretest was conducted in March-April, 2011 and post test was conducted in October-November, 2011.
  Fat percentage was measured using the bioimpedance machine InBody 720 and using skinfolds. Both registered body fat percentage.
Change from Baseline Cardiorespiratory fitness at 6 months | Data collected prior to (pre) and after (post) a 6 month intervention period. Pretest was conducted in March-April, 2011 and post test was conducted in October-November, 2011.
  Cardiorespiratory fitness was measure by a modified Balke protocol on a treadmill and registered in l/min.

SECONDARY OUTCOMES:
Age | This is one of the descriptive statistics which was collected at one time point only. Data were collected on day one, in april 2011.
  Age was assessed by questionaire to the nearest whole year.
Gender | This is one of the descriptive statistics which was collected at one time point only. Data were collected on day one, in april 2011
  Gender was assessed using a questionnaire and outcome was either Female or male.
Educational level | This is one of the descriptive statistics which was collected at one time point only. Data were collected on day one, in april 2011
  Educational level was assessed using a questionnaire as one of four different levels

OTHER OUTCOMES:
Physical activity level | This is one of the variables determining inclusion to the study and was collected at one time point only. Data were collected on day one, in april 2011
  Physical activity level was assessed using IPAQ- sf as minutes of physical activity per week.
Stage of change | This is one of the variables determining inclusion to the study and was collected at one time point only. Data were collected on day one, in april 2011
  Stage of change was assessed using a questionnaire as one of five alternatives.

CONTACTS AND LOCATIONS:
Overall Officials: Monica K Torstveit, PhD, Principal Investigator — University of Agder

IPD SHARING:
Plan to Share IPD: No
The IPD of the present study will be shared through publications (articles).

REFERENCES:
- [Derived] Kjaer IGH, Anderssen SA, Torstveit MK. A tailored telephone and email based exercise intervention induced reductions in various measures of body composition in physically inactive adults: A randomized controlled trial. Prev Med Rep. 2018 Jun 27;11:160-168. doi: 10.1016/j.pmedr.2018.06.011. eCollection 2018 Sep. PMID 29988751